CLINICAL TRIAL: NCT01725399
Title: Randomized Controlled Trial: Does First Oral Intake After Emergence From Anesthesia Predict the Incidence of Post-operative Vomiting in Children?
Brief Title: Does First Oral Intake After Emergence Predict the Incidence of Post-operative Vomiting in Children?
Acronym: XOndansetron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 12-1792
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Post-operative Vomiting
Keywords: post-operative vomiting
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water (Placebo Comparator): Water will be given as the study subject's first oral intake after emergence from general anesthesia.
  Interventions: Other: Water
- Apple Juice (Experimental): Apple juice will be given as the study subject's first oral intake after emergence from general anesthesia.
  Interventions: Other: Apple Juice

INTERVENTIONS:
Other: Apple Juice
  Arms: Apple Juice
Other: Water
  Arms: Water

SUMMARY:
Second only to pain, nausea and vomiting are the most uncomfortable complications of surgery and anesthesia. Unfortunately, our best defense against post-operative nausea and vomiting, a medicine called ondansetron (Zofran), is in dire national shortage. Consequently, non-pharmacological methods of prevention and treatment for post-operative nausea and vomiting have increased import. Following emergence from general anesthesia, children often request food and drink. There have been no studies to date that definitively determine the optimal first food or drink choice for these children. This study proposes to randomize children to either water or juice first intake following surgery. The investigators expect to find that children who consume glucose are less likely to vomit than those who first receive water.

ELIGIBILITY:
Inclusion Criteria:

* Dental surgery
* Tonsillectomy and adenoidectomy
* Strabismus surgery
* Age 2-18

Exclusion Criteria:

* Patient refusal
* Parent refusal
* Allergy / contraindication to ondansetron
* Prone to vomiting
* Inpatient
* Preoperative anxiolysis with ketamine
* Recovery location other than PACU
* Nil per os at baseline
* Presence of enteric tube
* Contraindication to any part of the study protocol

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Post-operative Vomiting | 24 hr post-op
  Patients will be assessed for vomiting upon entry to PACU until 24 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie R Wingate, MD, Principal Investigator — UNC Chapel Hill; Peggy P McNaull, MD, Study Chair — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States